CLINICAL TRIAL: NCT02170675
Title: Relative Bioavailability of Single Doses of 150 mg Dabigatran Etexilate (Capsule) When Administered Alone or in Combination With a Single Dose of 400 mg Ketoconazole (Tablet) or in Combination With 400 mg q.d. Ketoconazole (Tablet) at Steady State in Healthy Male and Female Volunteers (an Open Label, Fixed Sequence, Phase I Study)
Brief Title: Relative Bioavailability of Single Doses of Dabigatran Etexilate When Administered Alone or in Combination With a Single Dose of Ketoconazole or in Combination With q.d. Ketoconazole at Steady State in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.101
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Ketoconazole

ARMS (1):
- Dabigatran etexilate + Ketoconazole (Experimental): Period 1 - Dabigatran etexilate
  Period 2 - Dabigatran etexilate and single dose of 400 mg Ketoconazole on Day 8 and 9
  Period 3 - Dabigatran etexilate and multiple doses of 400 mg Ketoconazole on Day 10 to 16
  Interventions: Drug: Dabigatran etexilate; Drug: Ketoconazole

INTERVENTIONS:
Drug: Dabigatran etexilate
Drug: Ketoconazole

SUMMARY:
To investigate whether and to what extent the P-glycoprotein (P-gp) inhibitor ketoconazole affects plasma exposure of dabigatran.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥21 and ≤50 years
3. BMI range ≥18.5 and ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial, and intake of drugs which might reasonably influence the results of the trial within four weeks prior to administration or during the trial (e.g. P-gp inducers)
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
12. Alcohol abuse (more than 60 g/day)
13. Drug abuse
14. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
15. Excessive physical activities (within one week prior to administration or during the trial)
16. Any laboratory value outside the reference range that was of clinical relevance
17. Inability to comply with dietary regimen of trial site

    Exclusion criteria that were specific for this study:
18. Intake of medication, which influences the blood clotting, such as acetylsalicylic acid and oral vitamin K antagonists

    For female subjects:
19. Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
20. No adequate contraception during the study and until 1 month of study completion, i.e.

    implants, injectables, combined oral contraceptives, IUD [intrauterine device], sexual abstinence (for at least 1 month prior to enrolment), or surgical sterilisation (incl.

    hysterectomy). Females, who were not surgically sterile were asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)
21. Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for total dabigatran | up to Day 16
Maximum measured concentration of the analyte in plasma for total dabigatran | up to Day 16

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for free dabigatran | up to Day 16
Maximum measured concentration of the analyte in plasma for free dabigatran | up to Day 16
Maximum measured concentration of the analyte in plasma for dabigatran and BIBR 1087 SE, BIBR 951 BS | up to Day 16
Time from dosing to the maximum concentration of the analyte in plasma for dabigatran and BIBR 1087 SE, BIBR 951 BS | up to Day 16
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Area under the concentration-time curve of the analyte in plasma over the time interval from timepoints t1 to t2 for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 h for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Time from dosing to the maximum concentration of the analyte in plasma for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Terminal rate constant of the analyte in plasma for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Terminal half-life of the analyte in plasma for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Mean residence time of the analyte in the body after oral administration for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Apparent clearance of the analyte in the plasma after extravascular administration for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Apparent volume of distribution during the terminal phase λz following an extravascular dose for dabigatran | up to Day 16
  Dabigatran after each single dose (free and total after conjugate cleavage)
Changes from baseline in Vital signs (blood pressure [BP], pulse rate) | up to 14 days after last drug administration
Changes from baseline in 12-lead ECG | up to 14 days after last drug administration
Changes from baseline in Clinical laboratory tests (haematology, clinical chemistry, and urinalysis) | up to 14 days after last drug administration
Number of patients with adverse events | up to 14 days after last drug administration
Assessment of tolerability by the investigator | up to 14 days after last drug administration